CLINICAL TRIAL: NCT01494155
Title: Phase II Study of Neoadjuvant Accelerated Short Course Radiation Therapy With Proton or Photon RT Plus Capecitabine and Hydroxychloroquine for Resectable Pancreatic Cancer
Brief Title: Short Course Radiation Therapy With Proton or Photon Beam Capecitabine and Hydroxychloroquine for Resectable Pancreatic Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Theodore Sunki Hong, Radiation Oncologist, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 11-073
Record Dates: First submitted 2011-07-29; First posted 2011-12-16 (Estimated); Last update posted 2021-02-02 (Actual); Status verified 2021-02

CONDITIONS: Pancreatic Cancer
Keywords: resectable pancreatic cancer; pancreaticoduodenectomy
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Capecitabine; Hydroxychloroquine; Protons

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Hydroxychloroquine (Experimental): Hydroxychloroquine with chemoradiation
  Interventions: Drug: Capecitabine; Drug: Hydroxychloroquine; Radiation: Proton or Photon Radiation Therapy

INTERVENTIONS:
Drug: Capecitabine — 825 mg/m2 BID orally for a total of 10 days (M-F of weeks 2 and 3)
  Other Names: Xeloda
Drug: Hydroxychloroquine — 400 mg BID from study day 1 until surgery. Dosing resumed upon discharge from hospital
  Other Names: Plaquenil
Radiation: Proton or Photon Radiation Therapy — Daily, beginning Week 2 for 5 consecutive days

SUMMARY:
A standard treatment for patients with pancreatic cancer is standard photon radiation in combination with the chemotherapy drug, capecitabine. In this research study the investigators are using standard photon radiation or a different type of radiation therapy called proton beam radiation and adding hydroxychloroquine to be used in combination with capecitabine.

In this research study, the investigators are looking to determine if proton or photon beam radiation in combination with hydroxychloroquine and capecitabine is effective in controlling your cancer growth.

DETAILED DESCRIPTION:
Subjects will be treated in cycles of 28 days. Hydroxychloroquine will be taken orally, daily until the day before surgery and will resume after surgery until study end.

Capecitabine will be taken orally, daily. Proton or photon radiation treatment will start on Week 2 and will be delivered daily (5 days in a row, but not weekends or holidays). Radiation treatment will be give on an outpatient basis at the Francis H. Burr Proton Center or the Clark Center for Radiation Oncology at Massachusetts General Hospital.

The following tests will be performed weekly: physical exam, routine blood tests, optional blood tests and an eye exam every 3 months while taking hydroxychloroquine.

Subjects will have surgery (any time between Weeks 5 to 9) and after surgery resume taking hydroxychloroquine. Subjects will have a follow up visit every 3 months which will include: physical exam, routine blood tests, eye exam, and tumor assessment by chest and abdominal-pelvic CT scan or MRI (every 6 months for the first 2 years and yearly for years 3-5).

ELIGIBILITY:
Inclusion Criteria:

* Cytologic or histologic proof of pancreatic ductal carcinoma
* Life expectancy > 3 months
* Adequate organ and marrow function

Exclusion Criteria:

* Evidence of metastatic disease
* Pregnant or breast-feeding
* Tumors in the body or tail of the pancreas
* Serious concomitant systemic disorders such as significant cardiac or pulmonary morbidity (e.g. congestive heart failure, symptomatic coronary artery disease and cardiac arrhythmias not well controlled with medication) or myocardial infarction within the last 12 months, ongoing infection as manifest by fever
* Prior chemotherapy or radiation for treatment of the patient's pancreatic tumor
* Diagnosis of other invasive carcinomas (except basal cell carcinomas/squamous cell carcinoma of the skin) with the last 5 years. Carcinoma in-situ is allowed.
* Other serious uncontrolled medical conditions
* Lack of physical integrity of the upper gastrointestinal tract or malabsorption syndrome
* Known, existing uncontrolled coagulopathy
* Prior systemic fluoropyrimidine therapy (unless given in an adjuvant setting and completed at least 6 months earlier). Prior unanticipated severe reaction to fluoropyrimidine therapy, or known hypersensitivity to 5-fluorouracil or known DPD deficiency
* Participation in any investigational drug study within 4 weeks preceding the start of study treatment
* History of uncontrolled seizures, central nervous system disorders, or psychiatric disability
* Major surgery, excluding laparoscopy, within 4 weeks of the start of study treatment, without complete recovery
* Currently taking cimetidine
* Receiving any other study agents
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to capecitabine and HCQ
* Already taking HCQ or chloroquine for other diagnosis
* History of Grade 3 or greater retinopathy or keratitis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2011-12; Primary Completion 2022-01 (Estimated); Study Completion 2023-01 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival | 2 years
  To determine the progression-free survival of the addition of hydroxychloroquine to preoperative short course, chemoradiation therapy and adjuvant gemcitabine chemotherapy

SECONDARY OUTCOMES:
Pathologic response rate | 2 years
  To determine the complete pathologic response rate of preoperative capecitabine combined with hydroxychloroquine and short course radiation therapy in patients undergoing pancreaticoduodenectomy
Overall survival | 2 years
  To determine overall survival in patients treated with preoperative capecitabine + hydroxychloroquine and short course radiation therapy
Toxicity/Adverse events | 2 years
  To determine the toxicity of capecitabine + hydroxychloroquine and short course radiation therapy in patients with pancreatic cancer via analysis of frequency and grades of reported toxicities and adverse events, such as GI and hematologic toxicities, occurring in study participants
Surgical morbidity | 2 years
  To determine the surgical morbidity in patients undergoing pancreaticoduodenectomy who received preoperative capecitabine + hydroxychloroquine and external beam radiation therapy
Post-operative Mortality | 2 weeks
  To determine 30-day post-operative mortality after pancreaticoduodenectomy in patients who receive preoperative capecitabine and external beam radiation therapy
Biomarkers | 2 years
  To explore biomarkers of autophagy with hydroxychloroquine therapy and explore correlation with progression-free survival
Pathologic down-staging | 2 years
  To determine pathologic down-staging of hydroxychloroquine-based short course chemoradiation compared to a previous cohort (treated in prior study of neoadjuvant capecitabine + proton therapy)
Local control | 2 years
  To determine local tumor control at 2 years post treatment in study participants
Describe QoL | 2 Years
  To describe quality of life, symptom burden and mood in the study population
Measure utilization of health services | 2 years
  Measure utilization of health services (ER, hospital and ICU visits) in the study population

CONTACTS AND LOCATIONS:
Overall Officials: Theodore S Hong, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States